CLINICAL TRIAL: NCT00549445
Title: Effect of Macrolide Treatment on a Novel Pathway of Neutrophilic Inflammation in COPD
Brief Title: Effect of Macrolide Antibiotics on Airway Inflammation in People With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, J Edwin Blalock, Professor, Medicine-Pulm/Allergy/Clinical, University of Alabama at Birmingham
Other Study IDs: 1425; R01HL090999-01 (NIH); HL090999-01
Record Dates: First submitted 2007-10-24; First posted 2007-10-25 (Estimated); Results first posted 2017-08-14 (Actual); Last update posted 2017-09-29 (Actual); Status verified 2017-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Chronic Obstructive Pulmonary Disease; COPD; Exacerbation; Macrolide
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Azithromycin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Serum and Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Azithromycin-treated: Participants in the COPD Network Macrolide Study who received azithromycin for 1 year.
  Interventions: Drug: Azithromycin
- Placebo-treated: Participants in the COPD Network Macrolide Study who received placebo for 1 year.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azithromycin — 250 mg daily
  Groups: Azithromycin-treated
Drug: Placebo — Daily
  Groups: Placebo-treated

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a chronic lung disease. Azithromycin, an antibiotic, may be beneficial at reducing the symptoms and severity of the disease. This study will analyze previously collected study data to evaluate the anti-inflammatory properties of azithromycin and determine how azithromycin affects the frequency and severity of COPD exacerbations.

DETAILED DESCRIPTION:
COPD is a disease in which the lung airways are partly damaged and obstructed, making it difficult to breathe. The most common cause is cigarette smoking, but breathing in other types of lung irritants, including pollution, dust, and chemicals, over a long period of time may also contribute to COPD. It is the fourth leading cause of death in the United States. Symptoms include coughing, excess mucus production, shortness of breath, wheezing, and chest tightness.

Some bacterial infections may worsen COPD exacerbations. Current studies are examining if the macrolide antibiotic azithromycin may be beneficial at reducing the frequency and/or severity of COPD exacerbations. Azithromycin also has anti-inflammatory properties that may reduce the severity of COPD exacerbations by inhibiting the matrix metalloprotease (MMP)-catalyzed breakdown of collagen and the subsequent generation of proline-glycine-proline (PGP), a substance produced in response to collagen breakdown. An increase in PGP levels may indicate an increase in inflammation, which can worsen COPD symptoms. NHLBI's COPD Network Macrolide study includes people with COPD who were randomly assigned to receive either azithromycin or placebo for 1 year. For this current study, researchers will examine the Macrolide participants' previously collected blood samples, sputum samples, and study data, including information on COPD exacerbations and azithromycin effects. The purpose of this study is to examine the anti-inflammatory properties of azithromycin in people with COPD.

ELIGIBILITY:
Inclusion Criteria:

* Participating in the COPD Network Macrolide study
* Clinical diagnosis of at least moderate COPD
* Cigarette consumption of 10 pack years or more

Exclusion Criteria:

* Diagnosis of asthma
* Predicted life expectancy of less than 3 years
* History of hypersensitivity to macrolide antibiotics
* Long-term kidney insufficiency
* Long-term liver insufficiency
* Prolonged QT interval
* Use of medications that may prolong the QT interval

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2007-08; Primary Completion 2011-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James E. Blalock, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol Open to Accrual: August 2007, Primary Completion Date: July 2011 and Study Completion Date: July 2012. Recruitment location: University of Alabama at Birmingham and the Mayo Clinic.
Pre-assignment Details: This research was conducted as an ancillary study to a multicenter trial (NCT00325897) of the efficacy of azithromycin treatment for 1 year in preventing chronic obstructive pulmonary disease (COPD) exacerbations to test whether sputum levels of proline-glycine-proline (PGP) were altered by treatment or associated with exacerbation frequency.
Period: Overall Study
Arm/Group | Azithromycin-treated | Placebo-treated
Started | 23 | 30
Completed | 8 | 13
Not Completed | 15 | 17
Not completed — Sputum & Blood Samples Not Available | 15 | 17

BASELINE CHARACTERISTICS:
Population: The number of participants included in this study is small as sputum samples were available only from a minority of participants in the parent trial. Therefore, this greatly reduced the overall number of participants analyzed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Azithromycin-treated | Placebo-treated | Total
Number analyzed (Participants) | 23 | 30 | 53
Age, Continuous [Mean (Full Range); unit: years] | 64.4 [56 to 72.8] | 70.8 [62.4 to 79.2] | 67.6 [56 to 79.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 16
  Male | 17 | 20 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 12 | 23
  White | 12 | 18 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23 | 30 | 53

OUTCOME MEASURES:

1. Primary Outcome: Levels of PGP From Sputum Samples of COPD Patients Being Treated With Azithromycin.
Description: Nasopharyngeal swabs were obtained to determine if there is a reduction in PGP levels (including both PGP & Neutrophil-PGP) after chronic treatment with azithromycin.
  Unblinding of the parent trial revealed that there were 18 sputum samples from 13 placebo-treated participants and 14 sputum samples from 8 azithromycin-treated participants collected at months 1 through 12 of treatment (with sputum samples not being available, this greatly reduced the sample size).
Time Frame: Baseline to 12 months
Population: Levels of PGP from sputum samples are compared between subjects on the macrolide antibiotic, azithromycin, and subjects on placebo and correlated with neutrophil counts and protease activity in sputum.
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | Azithromycin-treated | Placebo-treated
Number analyzed (Participants) | 8 | 13
ng/mL | 2.27 [1.4 to 3.14] | 5.15 [3.61 to 6.69]
Statistical Analysis 1: Comparison: Azithromycin-treated vs Placebo-treated; Test type: Other — Student t test; p = 0.045, t-test, 1 sided — Threshold for significance is P-Value < 0.05

ADVERSE EVENTS:
Time Frame: From baseline to 12 months.
Description: This research was carried out as an ancillary study to the Macrolide trial of the NHLBI COPD Clinical Research Network (CRN). This was a prospective, parallel group, placebo-controlled, double-blind study of the efficacy of azithromycin in the chronic, outpatient management of COPD.
Arm/Group | Azithromycin-treated | Placebo-treated
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/13
Other Adverse Events (participants affected / at risk) | 0/8 | 0/13

LIMITATIONS AND CAVEATS:
We were limited by the number of participants included in this study is small, as sputum samples were available only from a minority of participants in the parent trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No